CLINICAL TRIAL: NCT07167147
Title: Survival Outcomes by Tumor-Node Stage and Recurrence Patterns in Colon Cancer After Radical Surgery
Acronym: STARS
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202500389B0
Record Dates: First submitted 2025-08-25; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Colon Cancer; Colon Adenocarcinoma; Colon Cancer Stage III; Colon Cancer Stage I; Colon Cancer Stage II; Cancer Recurrence; Survival Analysis
Keywords: Colon Cancer; Colon Adenocarcinoma; Stage I-III Colon Cancer; Tumor-Node Stage; TN Staging; Cancer Recurrence; Recurrence Patterns; Survival Outcomes; Radical Surgery; Prognostic Factors; Retrospective Cohort
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- T1-3N-: Patients with stage I-III colon adenocarcinoma, T1-3 tumors without lymph node involvement.
- T1-3N+: Patients with stage I-III colon adenocarcinoma, T1-3 tumors with lymph node involvement.
- T4N-: Patients with stage I-III colon adenocarcinoma, T4 tumors without lymph node involvement.
- T4N+: Patients with stage I-III colon adenocarcinoma, T4 tumors with lymph node involvement.

SUMMARY:
Colon cancer is one of the most common cancers worldwide, and even after curative (radical) surgery, some patients develop recurrence or distant metastasis. Understanding how tumor stage and lymph node status at the time of diagnosis influence the risk and patterns of recurrence is important for guiding follow-up and treatment strategies.

This study retrospectively evaluates patients with stage I-III colon cancer who underwent radical surgery at Chang Gung Memorial Hospital between 2006 and 2018. A total of 7,259 patients are included from the institutional tumor registry. Patients are categorized into four tumor-node (TN) stage groups:

* T1-3 without lymph node involvement
* T1-3 with lymph node involvement
* T4 without lymph node involvement
* T4 with lymph node involvement

The study aims to examine recurrence patterns (no recurrence, local recurrence, isolated lung metastasis, isolated liver metastasis, or multiple sites) and overall survival. Statistical analyses planned include Kaplan-Meier survival analysis and marginal structural models to compare outcomes across different TN stages and recurrence types.

This study is based on retrospective data and was approved by the Institutional Review Board of Chang Gung Memorial Hospital (IRB No: 202500389B0). No new patient enrollment or interventions will be performed, and patient consent was waived due to the retrospective nature of the study.

DETAILED DESCRIPTION:
Colon cancer remains a major cause of cancer-related morbidity and mortality worldwide. Even after curative resection, recurrence occurs in a significant proportion of patients, and survival outcomes vary depending on tumor and nodal status at diagnosis. While the TNM staging system is widely used for prognosis, the specific association between tumor-node (TN) combinations and recurrence patterns, as well as their impact on survival, is not fully established.

The objective of this study is to investigate the relationship between TN stage and recurrence patterns in patients with stage I-III colon adenocarcinoma who underwent radical surgery at Chang Gung Memorial Hospital, Taiwan. A retrospective cohort of 7,259 patients who had surgery between 2006 and 2018 is analyzed using data from the institutional tumor registry. Patients are categorized into four groups according to T and N status: T1-3N0, T1-3N+, T4N0, and T4N+.

Primary outcomes include recurrence patterns (local recurrence, isolated lung metastasis, isolated liver metastasis, multiple-site metastases, or no recurrence). The secondary outcome is overall survival, assessed both after surgery and after recurrence. Planned statistical analyses include multinomial logistic regression to evaluate recurrence risk by TN stage, Kaplan-Meier survival curves with log-rank tests to compare survival across recurrence types, and marginal structural models with inverse probability weighting to address time-dependent confounders and estimate causal effects of TN stage and recurrence on mortality risk.

This retrospective analysis was reviewed and approved by the Institutional Review Board of Chang Gung Memorial Hospital (IRB No: 202500389B0). Patient consent was waived because only de-identified registry data are used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed colon adenocarcinoma
* Stage I-III disease at diagnosis
* Underwent curative (radical) resection at Chang Gung Memorial Hospital between 2006 and 2018
* Availability of complete clinical, pathological, and follow-up data

Exclusion Criteria:

* Stage IV colon cancer at initial diagnosis
* Non-adenocarcinoma histology (e.g., undifferentiated carcinoma, squamous cell carcinoma, lymphoma, sarcoma)
* History of other malignancies or synchronous multiple cancers
* Patients who underwent only palliative surgery or local excision
* Incomplete medical records or missing follow-up information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included 7,259 patients with stage I-III colon adenocarcinoma who underwent curative resection at Chang Gung Memorial Hospital (Linkou, Taiwan) between 2006 and 2018. Patients were categorized into four groups according to tumor and nodal status: T1-3N-, T1-3N+, T4N-, and T4N+. Clinical, pathological, and survival data were collected from the institutional tumor registry for retrospective analysis.
Sampling Method: Non-Probability Sample
Enrollment: 7259 (Actual)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Recurrence Patterns After Radical Surgery in Stage I-III Colon Cancer | From date of radical surgery until the date of first documented recurrence, assessed up to 60 months.
  Recurrence classified as no recurrence, local recurrence, isolated lung metastasis, isolated liver metastasis, or multiple-site metastases, based on imaging and clinical follow-up data.
Overall Survival After Radical Surgery in Stage I-III Colon Cancer | From date of radical surgery until death from any cause, assessed up to 5 years.
  Defined as the time from surgery to death from any cause, assessed using hospital records and national death registry data.

SECONDARY OUTCOMES:
Disease-Free Survival | From date of radical surgery until the date of recurrence or death from any cause, whichever comes first, assessed up to 5 years.
  Time from surgery to first documented recurrence (local or distant) or death from any cause, whichever occurs first.
Cancer-Specific Survival (CSS) | From date of radical surgery until death specifically attributable to colon cancer, assessed up to 5 years.
  Time from surgery to death specifically attributable to colon cancer, assessed through clinical records and registry data.
All-Cause Mortality by Recurrence Pattern | From date of first documented recurrence until death from any cause, assessed up to 5 years.
  Mortality rates stratified by first recurrence type (local, isolated lung, isolated liver, multiple sites).
Prognostic Impact of Tumor-Node Stage | From date of diagnosis and radical surgery until the date of first documented recurrence or metastasis, assessed up to 5 years.
  Association between TN stage at diagnosis (T1-3N-, T1-3N+, T4N-, T4N+) and recurrence/metastasis risk, measured by multinomial regression models.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan District, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and ethical considerations. Only aggregated study results will be published in peer-reviewed journals.